CLINICAL TRIAL: NCT04617210
Title: Risk Factors for Postoperative Delirium in Elderly Patients Undergoing Major Non-Cardiac Surgery in Singapore
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/00117
Record Dates: First submitted 2020-10-30; First posted 2020-11-05 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Postoperative Delirium
Keywords: Geriatrics
MeSH Terms: conditions — Emergence Delirium | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical Cohort: Elderly patients aged 65 and above who are planned for major non-cardiac surgery predicted to be at least 2 hours in duration and requiring at least 1 postoperative stay in hospital.
  Interventions: Other: Neurocognitive tests and blood taking

INTERVENTIONS:
Other: Neurocognitive tests and blood taking — Battery of neurocognitive tests and questionnaires: MoCA, PHQ-9, Falls History, FIFE, STOPBANG, Nutritional Survey, CANTAB, Insomnia Severity Index, Bristol Activities of Daily Living Scale, NuDESC, 3D-CAM. Blood taking.

SUMMARY:
The primary aim is to establish the risk factors, in particular the modifiable risk factors, for the development of POD in elderly patients undergoing major non-cardiac surgery in a tertiary hospital in Singapore.

The secondary aims are:

1. To establish the incidence of POD in elderly patients in Singapore, including the proportions that develop hypoactive, hyperactive and mixed delirium, as well as dementia within a one-year follow-up period;
2. To understand the timeline of the development and peak incidence of POD, from the post-anaesthesia care unit till 3 days postoperatively;
3. To compare the utility and accuracy (sensitivity and specificity) of two simplified delirium detection tools, 3D CAM and NuDESC, against the gold standard DSM-5 criteria, in our population as a means for monitoring POD as standard of care in the future;
4. To collect data for holistic evaluation of neurobehavioural and daily functioning status

DETAILED DESCRIPTION:
Singapore's population is growing older and increasingly burdened with systemic disease. It is estimated that over 320 million people underwent surgery worldwide in 2010, with Asia being the fastest growing region. Elderly patients aged >65 years are presenting for surgery at an ever-increasing rate. In the United States, studies have estimated that approximately 53% of all surgical procedures are performed on patients over the age of 65. Projections estimate that approximately half of the population over the age of 65 will require surgery once in their lives.

We often hear from our elderly patients that they value their quality of life more than prolonging it. Therefore it is essential that we optimize the care in the perioperative period to allow patients to fully benefit from surgery, as this period profoundly impacts survival and quality of life of patients after surgery. There is a current focus on enhanced recovery after surgery (ERAS) where surgeons implement protocols such as improved analgesia, less invasive procedures and early mobilisation to encourage earlier discharge of post op patients. In the best practice guidelines for care of elderly surgical patients put forward by the American College of Surgeons National Surgical Quality Improvement Program (ACS NSQIP) and the American Geriatrics Society (AGS) published in 2012, anaesthesia plays a role in more than half of the 13 recommendations put forward.

One of these recommendations is to reduce postoperative delirium (POD). The anaesthetic agents we use is toxic to the brain, and deep anaesthesia causes POD, which is linked to increased hospital length of stay, increased 30-day mortality, and dementia. POD is one of the leading causes of why patients fall at home after surgery. Up to 10% will develop long-term neurocognitive deficits, which in turn diminish the quality of life and levy a tremendous socio-economic burden on family and care-givers, and shortens life. The topic of POD has dominated the anaesthesia literature in the last year, with both the US and European societies issuing best practice guidelines such as the Brain Health Initiative and the Safe Brain Initiative, as well as harmonization of the definitions of postoperative neurological outcomes with that used by neurologists in compliance with DSM-5 definitions to allow for collaborative solutions.

Awareness of POD remains poor amongst both doctors and the public. The reason for this is that POD requires specialized neurological testing and currently, there are no established biomarkers or monitors to detect it. Yet when patients are assessed for POD, it has been reported that it occurs in as many as 11-50% of patients undergoing major non-cardiac surgery. Studies have shown that up to 40% of POD is preventable. Anecdotally, POD is one of the leading reasons for in-hospital (blue letter) psychiatric referrals after surgery in NUHS, as delirious patients will refuse to comply with physiotherapy, medications and wound care, leading to delayed healing, infection and delayed discharge. Patients are not routinely assessed for POD, and can be discharged with it. Patients who are still delirious can end up with poor feeding and self-care, and even hurt themselves leading to rehospitalisation. In short, POD is a common yet under-diagnosed, and potentially preventable, complication of anaesthesia and surgery in the elderly that has significant long-term effects on the independence of patients after surgery and their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients aged 65 years and above
* Undergoing major non-cardiac surgery, defined as surgery that is predicted to be at least 2 hours and requiring at least 1 day postoperative stay in the hospital
* English, Chinese or Malay speaking

Exclusion Criteria:

* History of psychiatric disease
* Unable to provide informed consent for surgery
* Illiterate
* An active history of substance abuse
* Undergoing neurosurgical procedures
* Undergoing emergency surgeries
* Has a second surgery within 5 days of index surgery
* Non-resident of Singapore
* Severe hearing and/or speech impairment

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients aged 65 and above who are planned for major non-cardiac surgery predicted to be at least 2 hours in duration and requiring at least 1 postoperative stay in hospital.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-11-18 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Establish the risk factors for the development of POD in elderly patients undergoing major non-cardiac surgery in a tertiary hospital in Singapore. | Before surgery through to 1 year post surgery
  Collection of patient's demographics, medical records and surgical records to establish risk factors for POD development

CONTACTS AND LOCATIONS:
Overall Officials: Ne-Hooi Will Loh, Principal Investigator — National University Health System
Locations (1):
- National University Health System, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rose J, Weiser TG, Hider P, Wilson L, Gruen RL, Bickler SW. Estimated need for surgery worldwide based on prevalence of diseases: a modelling strategy for the WHO Global Health Estimate. Lancet Glob Health. 2015 Apr 27;3 Suppl 2(Suppl 2):S13-20. doi: 10.1016/S2214-109X(15)70087-2. PMID 25926315
- [Background] Yang R, Wolfson M, Lewis MC. Unique Aspects of the Elderly Surgical Population: An Anesthesiologist's Perspective. Geriatr Orthop Surg Rehabil. 2011 Mar;2(2):56-64. doi: 10.1177/2151458510394606. PMID 23569671
- [Background] Aldecoa C, Bettelli G, Bilotta F, Sanders RD, Audisio R, Borozdina A, Cherubini A, Jones C, Kehlet H, MacLullich A, Radtke F, Riese F, Slooter AJ, Veyckemans F, Kramer S, Neuner B, Weiss B, Spies CD. European Society of Anaesthesiology evidence-based and consensus-based guideline on postoperative delirium. Eur J Anaesthesiol. 2017 Apr;34(4):192-214. doi: 10.1097/EJA.0000000000000594. PMID 28187050
- [Background] Evered L, Silbert B, Knopman DS, Scott DA, DeKosky ST, Rasmussen LS, Oh ES, Crosby G, Berger M, Eckenhoff RG; Nomenclature Consensus Working Group. Recommendations for the nomenclature of cognitive change associated with anaesthesia and surgery-2018. Br J Anaesth. 2018 Nov;121(5):1005-1012. doi: 10.1016/j.bja.2017.11.087. Epub 2018 Jun 15. PMID 30336844